CLINICAL TRIAL: NCT01800253
Title: The Role of Acute Total Sleep Deprivation in the Regulation of Metabolism, Neuroendocrine Responses, and Behavioral Measures
Brief Title: The Effects of Acute Total Sleep Deprivation Versus Normal Sleep on Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SleepMetaJCCB2013
Record Dates: First submitted 2013-02-21; First posted 2013-02-27 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-11

CONDITIONS: Sleep Deprivation; Sleep
MeSH Terms: conditions — Sleep Deprivation | interventions — Blood Specimen Collection; Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total sleep deprivation (Experimental): Participants will be required to stay up for the entire night before 'Blood Samples' and 'Tissue samples' will be taken and the 'Portion Size Task' and 'Inhibitory task' will be performed. This will then be followed by the 'Oral glucose tolerance test' with additional 'Blood Samples' to be taken as described for that test.
  Interventions: Behavioral: Inhibitory task; Procedure: Blood samples; Procedure: Tissue samples; Procedure: Oral glucose tolerance test; Behavioral: Portion Size Task
- Sleep (Experimental): Participants will have an 8-h sleep opportunity before 'Blood Samples' and 'Tissue samples' will be taken and 'Portion Size Task' and 'Inhibitory task' will be performed. This will be followed by the 'Oral glucose tolerance test' with additional 'Blood Samples' to be taken as described for that test.
  Interventions: Behavioral: Inhibitory task; Procedure: Blood samples; Procedure: Tissue samples; Procedure: Oral glucose tolerance test; Behavioral: Portion Size Task

INTERVENTIONS:
Behavioral: Inhibitory task — Participants perform a binary decision on each presented stimuli. Of the two possible outcomes, participants are instructed to make a motor response (go) for one type, and are to withhold a response (no-go) for the other type. Reaction time and accuracy are measured for each event
Procedure: Blood samples — Hormone levels, neuromolecular levels and gene expression profiles will be analyzed from repeated blood samples obtained before and after the nighttime intervention
Procedure: Tissue samples — Expression profiles will be analyzed from samples obtained from tissues involved in metabolism
Procedure: Oral glucose tolerance test — 75 g of glucose will be dissolved in 300 ml of water and given to participants, followed by blood sampling at 0, 15, 30, 60, 90, 120 and 150 minutes following the ingestion of the glucose solution.
Behavioral: Portion Size Task — Participants are given a computer program that gives them the opportunity to choose the portions of a variety of food items that they would ideally like to consume

SUMMARY:
The study proposes to investigate whether acute total deprivation affects metabolism as measured through blood and peripheral tissues. Its aim is also to investigate how acute total sleep deprivation affects neurodegenerative markers, as well as hormones, memory performance and aspects of appetite regulation.

DETAILED DESCRIPTION:
It is predicted that acute total sleep deprivation will affect gene expression and DNA methylation. It is also predicted that sleep deprivation will up-regulate ghrelin, and affect other neuroendocrine markers and hormones in a negative manner. It is further predicted that sleep deprivation will decrease participants' memory performance.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 18-28y
* Healthy (self-reported) and not on medication
* Non-smoking
* Normal sleep-wake rhythm (i.e. 7-8 h per night, self-reported via diaries)

Exclusion Criteria:

* Major illness
* Taking any serious medications
* Any sleep conditions (e.g. irregular bedtimes, sleep complaints)
* Any dietary issues with the food items provided
* Current or history of endocrine, neurological or psychiatric disorders
* Shift work in the preceding three months or for a long duration
* Time travel over a significant number of time zones in the preceding two months
* Too much weight gain or weight loss in the preceding three months

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Gene expression and DNA methylation | Change from baseline (ie. around 1930 in the evening - before sleep intervention) to 12 hours later (around 0730 in the morning after the nighttime intervention), and to 15 hours later (around 1030 in the morning after the nighttime intervention)
  This study has been designed to measure the changes in gene expression and DNA methylation in circulating blood, i.e. mainly of white blood cells with active transcription and DNA regulation, and how this relates to possible changes in peripheral tissues involved in metabolism.

SECONDARY OUTCOMES:
Circulating hormone and neuromolecular levels | Change in circulating hormone levels from baseline (ie. around 1930 in the evening - before sleep intervention) to 12 hours later (around 0730 in the morning after the nighttime intervention)
  Participants will have their circulating hormone levels and neuromolecular levels taken and analyzed, including ghrelin, to determine if sleep deprivation alters hormone and neuromolecular levels related primarily to obesity, cognition or weight gain
Appetitive evaluation | Change in appetitive ratings after the sleep intervetion (from around 0700 in the morning after the nighttime intervention), repeated each hour
  Participants will be evaluated on their appetitive ratings in the morning following either nighttime intervention (acute total sleep deprivation or normal 8-hour sleep).
Portion Size Task | Change in selected portion size in the morning, at around 0830 hours in the morning following each nighttime intervention, and 2h30min later, i.e. 30 min after consuming an Oral glucose tolerance test, i.e. around 1100 hours
  Participants will be evaluated on their tendency to choose larger or smaller portions of a variety of meal items on a computer screen. This will be conducted both following partial sleep deprivation and normal sleep, and changes before and after glucose ingestion will be compared between these conditions
Inhibitory task | Change in cognitive inhibitory performance at around 0810 hours in the morning following the respective nighttime intervention.
  Participants perform a binary decision on each presented stimuli. Of the two possible outcomes, participants are instructed to make a motor response (go) for one type, and are to withhold a response (no-go) for the other type. Reaction time and accuracy are measured for each event.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Benedict, PhD, Principal Investigator — Department of Neuroscience, Uppsala University
Locations (1):
- Department of Neuroscience, Uppsala University, Uppsala, Uppsala County, Sweden

REFERENCES:
- [Derived] Zhang L, Grip A, Hjelmqvist D, Benedict C, Brandao LEM, Cedernaes J. Acute Sleep Loss Increases Circulating Morning Levels of Two MicroRNAs Implicated in Neurodegenerative Disease in Healthy Young Men. J Cell Mol Med. 2025 Apr;29(7):e70523. doi: 10.1111/jcmm.70523. PMID 40194981
- [Derived] Mateus Brandao LE, Espes D, Westholm JO, Martikainen T, Westerlund N, Lampola L, Popa A, Vogel H, Schurmann A, Dickson SL, Benedict C, Cedernaes J. Acute sleep loss alters circulating fibroblast growth factor 21 levels in humans: A randomised crossover trial. J Sleep Res. 2022 Apr;31(2):e13472. doi: 10.1111/jsr.13472. Epub 2021 Sep 2. PMID 34476847
- [Derived] Cedernaes J, Osler ME, Voisin S, Broman JE, Vogel H, Dickson SL, Zierath JR, Schioth HB, Benedict C. Acute Sleep Loss Induces Tissue-Specific Epigenetic and Transcriptional Alterations to Circadian Clock Genes in Men. J Clin Endocrinol Metab. 2015 Sep;100(9):E1255-61. doi: 10.1210/JC.2015-2284. Epub 2015 Jul 13. PMID 26168277